CLINICAL TRIAL: NCT01643161
Title: Guided Self-Help for Functional Neurological Symptoms: A Randomized Controlled Efficacy Trial
Brief Title: Guided Self-Help for Functional Neurological Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kari A. Martin, MD PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-005721
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Functional Neurologic Disease
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU+GSH (Experimental): Treatment As Usual plus Guided Self Help.
  Interventions: Behavioral: Treatment As Usual; Behavioral: Guided Self-Help
- TAU (Active Comparator): Treatment AS Usual.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Treatment As Usual — Communicating the diagnosis to the patient's primary care doctor and neurologist. May include referrals for physical therapy or psychiatric evaluations, or referrals to community therapists or doctors.
Behavioral: Guided Self-Help — A self-help workbook based on cognitive behavioral therapy, and four half-hour guidance sessions over a three-month period.
  Arms: TAU+GSH

SUMMARY:
Functional (psychogenic or somatoform) symptoms are commonly observed in neurology clinics. There is no known empirically validated treatment approach to functional symptoms. Cognitive Behavioral Therapy (CBT) can be effective, but there are major obstacles to its provision. The investigators will test the hypothesis that adding a CBT-based guided self-help (GSH) as compared to treatment as usual (TAU) improves patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult neurology outpatient with functional symptoms not largely explained by neurologic disease.

Exclusion Criteria:

* Unable to use the Guided Self-Help intervention, such as due to significant cognitive impairment or unable to comprehend English.
* Requires specialist psychiatric care.
* Has headache as the only symptom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
CGI | 3 months
  Clinical Global Improvement scale score (much worse, worse, same, better, much better) rated by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States